CLINICAL TRIAL: NCT06331351
Title: Effect of Jing Si Herbal Tea Liquid Packets on Chronic Pharyngolaryngitis: A Randomized, Double-blinded Clinical Trial
Brief Title: Effect of Jing Si Herbal Tea Liquid Packets on Chronic Pharyngolaryngitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dalin Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: A11203001-1
Record Dates: First submitted 2024-03-08; First posted 2024-03-26 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Chronic Pharyngitis
Keywords: Chronic pharyngitis; Jing Si herbal tea liquid packets; clinical trial
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): placebo: 2 times a day, 1 sachet each time.
  Interventions: Other: control group
- Jing Si herbal tea liquid packets group (Experimental): Jing Si herbal tea liquid packets: 2 times a day, 1 sachet each time.
  Interventions: Other: Jing Si herbal tea liquid packets

INTERVENTIONS:
Other: control group — 2 times a day, 1 sachet each time.
  Other Names: Placebo
  Arms: control group
Other: Jing Si herbal tea liquid packets — 2 times a day, 1 sachet each time.
  Arms: Jing Si herbal tea liquid packets group

SUMMARY:
Chronic pharyngolaryngitis is common and often make people suffer in many aspects. The etiology is numerous, for example, airway hypersensitivity, gastroesophageal acid regurgitation, sicca syndrome, anxiety, etc.

The investigators aimed to investigate the effect of Jing Si herbal tea liquid packets on chronic pharyngolaryngitis by a design of randomized, double-blind clinical trial in this study. The subjects who were bed-ridden, without self-care ability, receiving hemodialysis, no idea about the details of this study, poor compliance for this study, alcohol and/or drugs additives, pregnancy and breast-feeding women were excluded from this study.

A questionnaire for health and habits was performed at the start of the study, and a questionnaire for Reflux Symptom Index (RSI) was performed at the start and the end of the study. Finally, Student's t-test was used to test the difference between the Jing Si herbal tea group and the control group. And, multivariate linear regression was used to test the violation of clinical factors on the treatment outcome of Jing Si herbal tea liquid packets on chronic pharyngolaryngitis.

DETAILED DESCRIPTION:
Chronic pharyngolaryngitis is common and often make people suffer in many aspects. The etiology is numerous, for example, airway hypersensitivity, gastroesophageal acid regurgitation, sicca syndrome, anxiety, etc.

The investigators aimed to investigate the effect of Jing Si herbal tea liquid packets on chronic pharyngolaryngitis by a design of randomized, double-blind clinical trial in this study. One hundred and twenty adults of both sex with a range of age between of 20-70 years old were included. All participants were divided randomly into two groups. Jing Si herbal tea group received 1 pack of Jing Si herbal tea liquid packet twice a day for 1 month (30 days), and the control group received 1 pack of control liquid packet twice a day for 1 month (30 days). The subjects who were bed-ridden, without self-care ability, receiving hemodialysis, no idea about the details of this study, poor compliance for this study, alcohol and/or drugs additives, pregnancy and breast-feeding women were excluded from this study.

A questionnaire for health and habits was performed at the start of the study, and a questionnaire for Reflux Symptom Index (RSI) was performed at the start and the end of the study. Finally, Student's t-test was used to test the difference between the Jing Si herbal tea group and the control group. And, multivariate linear regression was used to test the violation of clinical factors on the treatment outcome of Jing Si herbal tea liquid packets on chronic pharyngolaryngitis.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women aged 20 to 70 years old.
2. Patients with chronic pharyngitis

Exclusion Criteria:

1. Patients who are bedridden or unable to take care of themselves.
2. Dialysis patients.
3. Patients who cannot understand the details of this study or cannot cooperate with the examination.
4. History of alcohol or drug abuse.
5. Pregnant and lactating women

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Health questionnaire | Before the test begins and after intervention completed (at 1 month)
  the recording items are as follows: age, gender, height, weight, waist circumference, disease history, smoking or not (quantification), drinking or not (quantification), and eating betel nut or not (quantification) , sleeping status, whether to drink coffee (quantification)
Reflux Symptom Index (RSI) | Before the test begins and after intervention completed (at 1 month)
  The Reflux Symptom Index (RSI) is in common use as a semi-quantitative tool to assess symptoms associated with laryngopharyngeal reflux (LPR).
  RSI is a scoring tool that consists of nine items used to assess various symptoms associated with LPR. Each item has a scale ranging from zero (no complaints) to five (severe complaints), with a maximum of 45 indicating the most severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Juen-Haur Hwang, MD, PhD, Study Chair — Dalin Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Locations (1):
- Dalin Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, Chiayi City, Taiwan

IPD SHARING:
Plan to Share IPD: No